CLINICAL TRIAL: NCT02724254
Title: A Double-blind Placebo Controlled, Randomized, Phase II Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Twice Daily Topical Applications of AP611074 5% Gel for up to 16 Weeks in Condyloma Patients
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Twice Daily Topical Applications of AP611074 5% Gel for up to 16 Weeks in Condyloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP611074.CT4
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Condyloma
Keywords: Genital warts; HPV types; Sexually Transmitted Disease; Papillomavirus Infections; Viral Disease; Anogenital warts; AGW; HPV6; HPV11; Human papillomavirus infection; HPV; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: conditions — Condylomata Acuminata; Sexually Transmitted Diseases; Papillomavirus Infections; Virus Diseases | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP611074 5% gel (Experimental): 100 mg twice daily doses of AP611074 5% gel
  Interventions: Drug: AP611074 5% gel
- Placebo (Placebo Comparator): AP611074 matching placebo gel
  Interventions: Drug: AP611074 matching placebo

INTERVENTIONS:
Drug: AP611074 5% gel
  Arms: AP611074 5% gel
Drug: AP611074 matching placebo
  Arms: Placebo

SUMMARY:
This is a double-blind placebo controlled, randomized, phase 2 study to assess the safety, tolerability, pharmacokinetics and efficacy of twice daily topical applications of AP611074 5% Gel for up to 16 weeks in condyloma patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged between 18 and 55 years.
2. External condylomas, 2-30 lesions (no more than 2 lesions side by side); flat or papular, but not pediculated.
3. Lesions must not be internal. Lesions that originate internally, but are visible externally will be considered internal and are not allowed in the study.
4. Total wart area (diameter x diameter) should not be less than 10mm2 and not more than 800 mm2
5. Individual wart area should not measure more than 50mm2, and the major perpendicular diameter should not measure more than 10mm (1cm).
6. Lesions to be treated should have appeared between 1 to 6 months before screening, and patients should not have received any previous condyloma treatment during the last 2 months before enrollment.
7. For female patients: either postmenopausal, taking adequate contraceptive method or surgically sterile.

Exclusion Criteria:

1. Patients should not have received genital wart treatment for previous condylomas (other than the prior treatment for current condylomas referred at inclusion criteria) in the last 12 months before enrollment
2. Patients with any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease, transplanted or immunosuppressed patients or other clinical condition that, in the Investigator's judgment, prevents the patients from participating to the study.
3. Patients with any clinically significant abnormality following review of screening laboratory tests, vital signs, full physical examination and ECG.
4. Patients with history or presence of drug or alcohol abuse.
5. Patients with positive HBs or HBc antigen or anti HCV antibody, or positive results for HIV 1 or 2 tests.
6. Patients using any dermatological drug therapy in the treatment area during the last month prior the first application of the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one local skin reaction (LSR) | Day 0 to Week 16
Number of patients experiencing adverse events | Day 0 to Week 16
Mean plasma concentrations of AP611074-04 | Day 0 to 2 weeks post end of treatment

SECONDARY OUTCOMES:
Proportion of subjects with a complete clearance rate (100%) for baseline genital wart lesions | Day 0 to week 16
Reduction in the total condyloma area for lesions | Day 0 to week 16
Proportion of subjects with a complete clearance rate (100%) for all genital wart lesions | Day 0 to week 16
Time to complete clearance | Day 0 to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Aviragen Therapeutics, Inc.
Locations (12):
- Argentina (5):
  - Anaconda Invesigational Site, Buenos Aires
  - Anaconda Investigational Site, Buenos Aires
  - Anaconda Investigational Site, Córdoba
  - Anaconda Investigational Site, Mendoza
  - Anaconda Investigational Site, Sante Fe
- Chile (2):
  - Anaconda Investigational Site, Concepción
  - Anaconda Investigational Site, Santiago
- Ecuador (3):
  - Anaconda Investigational Site, Cumbayá
  - Anaconda Investigational Site, Guayaquil
  - Anaconda Investigational Site, Quito
- Serbia (2):
  - Anaconda Investigational Site, Belgrade
  - Anaconda Investigational Site, Novi Sad